CLINICAL TRIAL: NCT03072758
Title: Men's Club: Impact of Male Partner Involvement on Initiation and Sustainment of Exclusive Breastfeeding Among Postpartum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: University Of Nigeria Teaching Hospital (Network); Catholic Caritas Foundation, Nigeria (Unknown)
Responsible Party: Principal Investigator, Echezona Ezeanolue, Professor of Public Health and Pediatrics, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 959559-3
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: HIV Infections; Breastfeeding, Exclusive
Keywords: Male partner involvement
MeSH Terms: conditions — HIV Infections; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men's Club Intervention Group (Experimental): Participants randomized to this group will receive interventions from the study team.
  Interventions: Behavioral: Men's Club
- Men's Club Control Group (No Intervention): Male participants in the control group will receive only education pamphlets related to breastfeeding during the 3rd trimester of their female partner's pregnancy

INTERVENTIONS:
Behavioral: Men's Club — Interactive session: This will be a one-day five-hour session that will take place at the church, and will be facilitated by trained lactation nurses. This will involve a maximum of 10 male participants and will occur during the female partner's 3rd trimester. Male partners will (a) complete a structured questionnaire to determine baseline knowledge, attitudes and beliefs about breastfeeding practices, and (b) actively engage in educational information on the benefit of exclusive breastfeeding. At the end of the session, the participants will receive educational pamphlets on breastfeeding to reinforce all the information that had been provided.
  Phone call reminders: Participants will receive weekly robocalls during the first six weeks following the birth of the infant to reinforce the benefits of exclusive breastfeeding. This will be an automated service that will deliver the calls at a specific time of the day the participants have indicated on their questionnaire.
  Arms: Men's Club Intervention Group

SUMMARY:
Breastfeeding remains the optimal mode of feeding for infants younger than six months. Exclusive Breast Feeding (EBF) among HIV-infected mothers has been shown to be associated with a sustained and significant reduction in HIV transmission and has the potential to reduce infant and under-five mortality.

Given the considerable authority among men as decision makers in sub-Saharan African, we may be witnessing a missed opportunity to engage men in the education, awareness, and decision-making for EBF. Understanding the role and impact of male partners on this decision-making process require further examination to inform the development of effective and sustainable evidence-based interventions to support the initiation and sustainment of EBF.

DETAILED DESCRIPTION:
Summary of the Parent Grant (R01HD087994): The parent grant is a cluster randomized comparative effectiveness trial designed to test the effectiveness of an integrated intervention for sustained testing and retention (iSTAR) on linkage, engagement, and retention among women with HIV infection. The iSTAR intervention provides: confidential, onsite integrated laboratory testing during baby showers; a network of church-based health advisors; clinic based teams trained in motivational interviewing; quality improvement skills to engage and support HIV-infected women; and integrated case management to reduce loss to follow-up. Primary outcomes are the difference in linkage and engagement rates between iSTAR and the clinic-based control group (CG). The secondary outcomes are the difference in retention and viral suppression rate.

Building upon the parent grant, this administrative supplement grant will assess the comparative effectiveness of Men's Club (MC) as intervention group (MC-IG) compared to the control group (MC-CG) on the initiation and sustainment of exclusive breastfeeding. Men's Club is an integrated intervention where male participants receive a five-hour interactive/educational session during their partner's pregnancy, and weekly phone reminders during the first six-week postnatal period to increase EBF knowledge and support strategies, and to improve sustainment of EBF respectively. Male partners in MC-CG will not receive the proposed intervention. Additionally, we will explore barriers and facilitators to support and sustainment of exclusive breastfeeding among participants from both MC-IG and MC-CG in the study. The Primary Outcome is the difference in the rate of initiation and sustainment of EBF between the two groups. The Secondary Outcome is the difference in knowledge of feeding options among male partners and rate of sustained EBF among the female partners in the two groups at 6 months post-delivery.

ELIGIBILITY:
Inclusion Criteria:

* Cohabiting couples/partners; residing in Benue state, Nigeria identified during iSTAR recruitment (baby showers)

Exclusion Criteria:

* HIV-infected females who have not disclosed their status to their male partners; male partners who do not own a phone; multiple pregnancy; and any health-related condition that prevents the female partner from breastfeeding.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Initiation of breastfeeding | 6 weeks
  Provision of mother's breast milk to infants within one hour of birth; participant self-report during face-to-face interview at 6 weeks post-partum
Sustainment of exclusive breastfeeding | 3 months
  Any/exclusive breastfeeding at 3 months is measured using a structured questionnaire at 3 months postnatal
Difference in rates of sustainment of exclusive breastfeeding | 6 months
  Any/exclusive breastfeeding at 6 months is measured using a structured questionnaire at 6 months postnatal

SECONDARY OUTCOMES:
Difference in breastfeeding knowledge | Baseline and 6 weeks
  Breastfeeding Knowledge Questionnaire (survey) at prenatal timepoint and 6 weeks postpartum
Attitudes towards breastfeeding | 6 weeks
  Iowa Infant Feeding Attitudes Scale (survey) at 6-weeks post delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Caritas Foundation, Makurdi, Benue State, Nigeria

IPD SHARING:
Plan to Share IPD: No